CLINICAL TRIAL: NCT01411085
Title: Alcoholism and Schizophrenia: A Translational Approach to Treatment
Brief Title: Risperidone and Desipramine in Alcohol Use and Schizophrenia
Acronym: RADIAUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: University of South Carolina (Other); University of Massachusetts, Worcester (Other); Michigan State University (Other)
Responsible Party: Principal Investigator, Alan Green, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R21AA019534-01A1 (NIH)
Record Dates: First submitted 2011-06-16; First posted 2011-08-08 (Estimated); Results first posted 2018-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Schizophrenia; Alcoholism; Dual Diagnosis
Keywords: Schizophrenia; Alcoholism; Dual Diagnosis; Desipramine; Risperidone
MeSH Terms: conditions — Schizophrenia; Alcoholism | interventions — Risperidone; Desipramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Risperidone + Desipramine (Experimental): All participants will be treated with risperidone (or a risperidone-like agent including: risperidone long-acting, paliperdione, and paliperidone palmitate) at the time treatment with desipramine is initiated. The target dose of oral risperidone is 4mg though variations are allowed. The target dose of desipramine is 100mg.
  Interventions: Drug: Risperidone + Desipramine

INTERVENTIONS:
Drug: Risperidone + Desipramine
  Other Names: Norpramin

SUMMARY:
Note: In June 2013, the study design was changed from a randomized controlled study of risperidone + despiramine vs. risperidone vs. placebo to an open label pre-post study of risperidone (or risperidone-like drug) + desipramine. The aims of the study were revised to read:

1. To determine whether participants treated with risperidone in combination with desiprmaine have less alcohol use (fewer drinking days; fewer heavy drinking days) during the final 8 weeks on these medications as compared to pre-baseline. The primary hypothesis is that compared to pre-baseline, participants will demonstrate fewer days of drinking (per week), as well as fewer days of heavy drinking (per week) in the final eight weeks they are taking risperidone and desipramine, as recorded on the Timeline Follow-Back assessment
2. To explore changes in symptoms (of schizophrenia and of depression) in the final eight weeks of treatment with risperidone + desipramine compared to the period before baseline
3. To assess the side effect burden associated with the combination of these two medications in participants.

The original aims of the study were:

The purpose of this study is to determine whether participants who are treated with risperidone in combination with desipramine have less alcohol use (fewer drinking days; fewer heavy drinking days) than do participants who are treated with RISP with placebo. The primary hypothesis is that compared to treatment with risperidone, participants randomized to a combination of risperidone plus desipramine will have fewer days of drinking, as well as fewer days of heavy drinking. The study will also compare the effects of risperidone as compared to risperidone plus desipramine on participants' symptoms and side effects.

DETAILED DESCRIPTION:
Alcohol use disorder is at least three times more common in schizophrenia than in the general population, and worsens the course of schizophrenia. Typical antipsychotic agents are of limited value in controlling alcohol use in these "dual diagnosis" patients. Data from our group and others suggest that the atypical antipsychotic drug clozapine limits alcohol and cannabis use in "dual diagnosis" patients with schizophrenia much more effectively than other antipsychotics that have been assessed, however, the side effects produced by clozapine severely limit its use.

The investigators have hypothesized that clozapine will lessen alcohol/substance use in such dual diagnosis patients in part because of its mechanism of action that includes release of dopamine (DA) in the prefrontal cortex which will help to normalize dysfunctional brain reward circuits that may underlie the co- occurring alcohol/substance use in patients with schizophrenia. Our data suggest that the effect of clozapine can be duplicated in rodents when medications with clozapine-like activity (DA D2 antagonism, potent norepinephrine (NE) α2 receptor antagonism and NE reuptake inhibition) are combined together. The investigators have demonstrated that RISP (a medication that is both a DA D2 receptor antagonist, and a potent NE α2 receptor antagonist), in combination with the specific NE reuptake inhibitor desipramine, significantly decreases alcohol consumption in alcohol drinking rodents.

This translational study is a pilot "proof of concept" 14-week double-blind investigation of participants who have co-occurring diagnoses of schizophrenia and an alcohol use disorder. Patients not treated with risperidone (or a risperidone-like agent, including risperidone long-acting, paliperidone and paliperidone palmitate) at the time of consent will be switched to oral risperidone in the first two weeks of the study. At Week 3, all participants will begin treatment with risperidone risperidone plus desipramine and followed for 12 weeks. The primary outcome measure will be days of drinking (per week), as well as days of heavy drinking (per week). The investigators anticipate that data from this study will support a larger trial of risperidone + desipramine in patients with schizophrenia and an alcohol use disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the diagnostic criteria of schizophrenia or schizoaffective disorder
2. Meets the diagnostic criteria for a current alcohol use disorder (abuse or dependence)
3. Recent alcohol use as documented on the Timeline Followback
4. Receives outpatient treatment with oral antipsychotic medication (including risperidone.
5. Is willing to switch to risperidone treatment at the beginning of the study.

Exclusion Criteria:

1. Other substance use disorder other than alcohol, caffeine and nicotine, and cannabis abuse, as defined by DSM-IV criteria.
2. Receives current treatment with Clozapine
3. Continues to use alcohol despite current adequate treatment with medication to decrease alcohol use(e.g. naltrexone, acamprosate, disulfiram or topiramate)
4. Is determined to be a "slow metabolizer" of CYP2D6
5. Is currently pregnant, trying to become pregnant, or nursing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-12; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan I Green, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (4):
- United States (4):
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Michigan State University / Cherry Street Health Services, Grand Rapids, Michigan
  - Dartmouth Medical School, Lebanon, New Hampshire
  - University of South Carolina School of Medicine, Columbia, South Carolina

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants were enrolled in a risperidone + placebo arm, but in 6/2013 the design of the study was changed to include only the risperidone + desipramine arm.
Groups:
- Risperidone + Desipramine: All participants were treated with risperidone (or risperidone-like agent, including risperidone long-acting, paliperidone and paliperidone palmitate) at the time that treatment with desipramine was initiated. The target of oral risperidone was 4 mg/day, though variations were allowed. The target dose of desipramine was 100 mg/day.
Period: Overall Study
Arm/Group | Risperidone + Desipramine
Started | 10
Completed | 7
Not Completed | 3
Not completed — Physician Decision | 1
Not completed — Protocol Violation | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: 7 completers in the risperidone + desipramine group were analyzed. 3 study subjects in the risperidone + desipramine group did not have sufficient days in study for analysis.
Groups:
- Risperidone + Desipramine: All participants were treated with risperidone (or risperidone-like agent, including risperidone long-acting, paliperidone or paliperidone palmitate) at the time treatment with desipramine was initiated. The target dose of oral risperidone was 4 mg/day, though variations were allowed. The target dose of desipramine was 100 mg/day.
Arm/Group | Risperidone + Desipramine
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants] — Population: 10 study subjects were enrolled.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 10
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 10 study subjects were enrolled.
  years | 46 (9.82)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 10 study subjects were enrolled.
  Participants
    Female | 1
    Male | 9
Region of Enrollment [Count of Participants; unit: Participants] — Timeline Followback assessment of drinks per week Population: 10 study subjects were enrolled.
  Participants
    United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Timeline Followback Assessing Number of Drinks Per Week
Description: Alcohol/other substance use (including tobacco) will be assessed primarily by weekly self-report using the Timeline Followback (TLFB) method enhanced by procedures to strengthen the reliability and validity of this measure. It involves asking participants to retrospectively estimate their alcohol and other substance use.
Time Frame: Weekly for 14 weeks, using data from last 8 weeks
Population: The analysis was performed on all completers (N=7).
Measure: Mean (Standard Deviation); unit: Drinks per week
Groups:
- Risperidone + Desipramine: All participants were treated with risperidone (or a risperidone-like agent, including risperidone long-acting, paliperidone or paliperidone palmitate). The target dose of oral risperidone was 4 mg/day, though variations were allowed. The target dose of desipramine was 100 mg/day.
Arm/Group | Risperidone + Desipramine
Number analyzed (Participants) | 7
Drinks per week | 35.9 (20.4)
Statistical Analysis 1: Comparison: Risperidone + Desipramine; The assessment was between baseline and values for last 8 weeks; Test type: Superiority; p = 0.317, t-test, 2 sided; Mean Difference (Final Values) = 7.0

ADVERSE EVENTS:
Groups:
- Risperidone + Desipramine: All participants were treated with risperidone (or a risperidone-like agent including: risperidone long-acting, paliperdione, and paliperidone palmitate) at the time treatment with desipramine is initiated. The target dose of oral risperidone is 4mg/day though variations were allowed. The target dose of desipramine was 100mg/day.
  Risperidone + Desipramine
Arm/Group | Risperidone + Desipramine
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risperidone + Desipramine (N=10)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Suicide atttempt (Psychiatric disorders) | 1 (1)
Alcohol intoxication (Psychiatric disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risperidone + Desipramine (N=10)
Anxiety (Psychiatric disorders) | 1 (2)
Depression (Psychiatric disorders) | 1 (1)
Diarrehea (Gastrointestinal disorders) | 1 (1)
Dizziness (General disorders) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Gum Infection (Infections and infestations) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Increased appetite (Gastrointestinal disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Irritability (General disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Libido decrease (Psychiatric disorders) | 1 (1)
Involuntary movements (Nervous system disorders) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Abnormal ECG (Investigations) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 4 (6)
Right bundle branch (Cardiac disorders) | 1 (1)
Alcohol intoxication (Psychiatric disorders) | 1 (7)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 2 (3)
Tachycardia (Cardiac disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1)
GERD (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No